CLINICAL TRIAL: NCT00787111
Title: Extended Management & Measurement of Autism (Emma): An Open-Label, Follow-On Study to Investigate the Safety and Impact on Developmental Trajectory of 18 Months Treatment With Fluoxetine Orally Dissolving Tablet (Odt) In Childhood and Adolescent Autistic Disorder
Brief Title: Extended Management and Measurement of Autism
Acronym: EMMA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Neuropharm (Industry)
Collaborators: Autism Speaks (Other)
Responsible Party: Dr. Mike Snape/ Chief Scientific Officer, Neuropharm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPL-2008-4-AUTUS-005
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Autistic Disorder
Keywords: Drug: Fluoxetine
MeSH Terms: conditions — Autistic Disorder | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoxetine ODT (Experimental): Fluoxetine ODT ranging from 2mg to 54mg
  Interventions: Drug: Fluoxetine (prozac)

INTERVENTIONS:
Drug: Fluoxetine (prozac) — Formulation: ODT

SUMMARY:
This open-label research study will continue to monitor the safety of fluoxetine in children after their completion of a previous double-blind placebo controlled clinical study, with fluoxetine. The study will also look at the effect of fluoxetine on IQ (Intelligence Quotient) over an 18 month period.

DETAILED DESCRIPTION:
This research study will monitor the safety of fluoxetine in all patients after their completion of the previous clinical study, in which they received fluoxetine or placebo. The study will look at the effect of fluoxetine on IQ (Intelligence Quotient) over an 18 month period. A possible total of 128 children and adolescents with AD will participate in the study from sites across the US.

The study is open-label. All of the subjects in this study will receive the active medicine fluoxetine orally dissolving tablets (ODT). Children will begin by receiving a daily dose of 2mg fluoxetine for two weeks. The family and child will be asked to come back to the clinic 2 weeks later and, depending on the child's tolerance and response to the medicine, may have his or her dose increased to 4mg/day. After this visit, the time between visits to the clinic and the dose that the child will receive will be decided by the study investigator based on their clinical judgment on benefit versus tolerability. The largest daily dose of fluoxetine that the child could receive in this study is 54mg.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have met the inclusion criteria for the preceding double-blind SOFIA Study, and must have completed at least 10 weeks of treatment in the 14 week SOFIA study or have withdrawn from the SOFIA study due to worsening of clinical symptoms (i.e. a CGI-I-AD of 6 or 7 which, in the Investigator's opinion, required alternative intervention except symptoms of activation which could not be ameliorated by reduction in dose).
2. Patients must have been free of fluoxetine and other SSRI's for 4 weeks prior to the first dose of open-label medication (washout).
3. Female patients who have reached menarche must have a negative pregnancy test at baseline and as required, in the opinion of the Investigator.
4. Females of childbearing potential must be using a medically accepted means of contraception not affected by fluoxetine treatment, or must remain abstinent for the duration of the study.
5. Patients must be able to follow the Investigator's instructions and be able to comply with visit requirements
6. Each Legally Authorized Representative (usually parent or guardian) must have a level of understanding sufficient to provide written informed consent to all required tests and procedures.
7. As required by the local or central IRB, the patient should assent to all required tests and procedures.

Exclusion Criteria:

1. Patients who experienced a serious adverse event during the double-blind SOFIA Study which was determined to be related to the study medication by the Investigator or the sponsor
2. Patients who were unable to tolerate the lowest dose of study medication in the double-blind SOFIA study (2mg fluoxetine or placebo) should not be enrolled in this study
3. Diagnosis of Rett Syndrome, Childhood Disintegrative Disorder
4. Patients currently taking psychotropic medication are excluded. Patients can be enrolled in the study if the psychotropic medication has been completely withdrawn prior to the baseline visit; for at least two weeks for neuroleptics / atypical antipsychotics and for at least 5 days for stimulants
5. Patients exhibiting high levels of aggression, irritability or self injurious behavior to the extent that in the Investigator's opinion the patient would be more appropriately treated with psychotropic medication other than fluoxetine such as an atypical antipsychotic
6. Patients currently taking a monoamine oxidase inhibitor. Patients who have stopped taking an irreversible MAOI should be free of medication for at least 2 weeks prior to the baseline visit and medication free for at least one day after stopping a reversible MAOI A.
7. Patients with diabetes who are treated with insulin
8. Patients currently taking tramadol, triptans (e.g.sumatriptan), lithium, tryptophan, haloperidol, clozapine, flecainide or encainide, vinblastine, carbamazepine, tricyclic antidepressants, phenytoin or warfarin are also excluded from the study.
9. Current treatment with the herbal remedy, St John's Wort (Hypericum perforatum)
10. History of, or current cardiovascular, renal, hepatic, respiratory and particularly gastrointestinal disease which may interfere with the absorption, distribution, metabolism or excretion of the study medication.
11. History of, or current cerebrovascular disease or brain trauma.
12. History of, or current significant endocrine disorder, e.g. hypo or hyperthyroidism.
13. History of or current malignancy.
14. Presence of psychotic symptoms or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder, as assessed by the Investigator.
15. Judged clinically to be at risk of suicide (suicidal ideation, severe depression, or other factors), as assessed by the Investigator.
16. Current active seizure disorder
17. Tourette's Disorder.
18. Female patients who are either pregnant or nursing.
19. Documented history of hypersensitivity or intolerance to SSRIs
20. Current drug abuse or dependence disorder or dependency in the 3 months prior to the baseline visit.
21. Clinically significant abnormalities in safety laboratory tests or vital signs as measured at baseline (as applicable) that would put the patient at substantially increased risk from study medication

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Safety Outcomes: Laboratory determinations, Urine drugs of abuse tests,Vital Signs,Physical Examinations, Adverse Events/Serious Adverse Events, Clinical Global Impression of Severity (CGI-S AD) | through the study

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Southwest Autism Research and Resource Centre, Phoenix, Arizona
  - University of California Davis, Sacramento, California
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - University of Illinois, Chicago, Illinois
  - AMR-Baber Research Inc., Naperville, Illinois
  - Harvard Medical School, Medford, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - CRCNJ, Voorhees Township, New Jersey
  - Long Island Jewish Hospital, Bethpage, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio
  - Seattle Children's Hosptial University of Washington, Seattle, Washington